CLINICAL TRIAL: NCT00998465
Title: Hemodynamics, Salt Sensitivity and Body Composition in Patients With Morbid Obesity - Effect of Weight Loss Following Laparoscopic Gastric Bypass
Brief Title: Hemodynamics, Salt Sensitivity and Body Composition in Patients With Morbid Obesity
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Peter Kramshoj Bonfils, MD, University Hospital Koege
Other Study IDs: SJ-99
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Obesity; Hypertension
Keywords: Obesity; Hypertension; Salt sensitivity; Laparoscopic gastric bypass; Bariatric surgery
MeSH Terms: conditions — Obesity; Hypertension | interventions — Blood Pressure; Absorptiometry, Photon; Plasma Volume; Glomerular Filtration Rate; Blood Specimen Collection; Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples: p-glucose, p-insulin, MR-proANP, hemoglobine, sodium, potassium, creatinine, albumine.
  Urine collections: u-sodium, u-potassium, u-creatinine

GROUPS / COHORTS (3):
- Obese, hypertension: Obese patients with hypertension and a body mass index 40-50 kg/m2
  Interventions: Other: 24-hour blood pressure; Other: Echocardiography; Other: Inert gas rebreathing; Radiation: Dexa-scan; Radiation: Plasma volume; Radiation: Glomerular filtration rate (GFR); Other: Blood samples; Other: Urine analyses; Dietary Supplement: Diets with low and high sodium content
- Control: Control subjects without hypertension and body mass index < 30 kg/m2
  Interventions: Other: 24-hour blood pressure; Other: Echocardiography; Other: Inert gas rebreathing; Radiation: Dexa-scan; Radiation: Plasma volume; Radiation: Glomerular filtration rate (GFR); Other: Blood samples; Other: Urine analyses; Dietary Supplement: Diets with low and high sodium content
- Obese, normotension: Obese patients without hypertension and a BMI between 40-50 kg/m2
  Interventions: Other: 24-hour blood pressure; Other: Echocardiography; Other: Inert gas rebreathing; Radiation: Dexa-scan; Radiation: Plasma volume; Radiation: Glomerular filtration rate (GFR); Other: Blood samples; Other: Urine analyses; Dietary Supplement: Diets with low and high sodium content

INTERVENTIONS:
Other: 24-hour blood pressure — Blood pressure is measured every 15 minutes in the daytime and every 30 minutes at night
Other: Echocardiography — Standard 2-D and m-mode echocardiography with determination of dimensions, systolic, and diastolic function.
Other: Inert gas rebreathing — Cardiac output, stroke volume and total peripheral resistance are tested at rest and during exercise (bicycle ergometer) using non-invasive equipment (inert gas rebreathing - Innocor)
Radiation: Dexa-scan — Fat mass and fat free mass is determined with a whole body Dexa scan, and bone mineral density is tested with Dexa-scans of the lumbar spine and proximal femur.
Radiation: Plasma volume — The test is performed using 5 MBq technetium-labeled albumine (99mTc-albumine - Vasculosis) with several postinjection samples for accurate zero-time extrapolation.
Radiation: Glomerular filtration rate (GFR) — GFR and ECV are determined following injection of 3,7 MBq 51Cr-EDTA and postinjection samples three-four hours after injection.
Other: Blood samples — p-glucose, p-insulin, NT-proBNP, hemoglobin, potassium, sodium, creatinine, albumine
Other: Urine analyses — 24-hour urine collections with determination of u-sodium, u-potassium and u-creatinine.
Dietary Supplement: Diets with low and high sodium content — Participants are subjected to 5 days of low (90 mmol/day) and high (250 mmol/day) sodium intake in a randomized order before and 1 year after laparoscopic gastric bypass surgery.

SUMMARY:
The purpose of this study is to evaluate the effect of high vs. low sodium intake on blood pressure and system hemodynamics in patients with morbid obesity and to evaluate the impact of laparoscopic gastric bypass on blood pressure, salt sensitivity and body composition in morbidly obese patients. Furthermore, we wants to describe the hemodynamic mechanisms involved in the amelioration of blood pressure during long-term weight loss.

DETAILED DESCRIPTION:
Overweight and obesity are rapidly increasing in Western countries and are associated with increased mortality and morbidity. The increased morbidity is assumed to be mediated mainly by insulin resistance, diabetes, hypertension and lipid disturbances, but obesity also represents an independent risk factor for cardiovascular disease.

Obesity is associated with an increased risk of hypertension but the pathophysiological basis is not fully established. Several studies have indicated that blood pressure of obese patients could be more dependent on dietary sodium intake than the blood pressure of non-obese patients(as it is the case for patients with essential hypertension)and that this sodium sensitivity of blood pressure is lost after weight loss.

To date, bariatric surgery is the only therapy resulting in substantial and durable long-term weight loss, and the beneficial effects on obesity-related co-morbidities have been well documented. Laparoscopic gastric bypass results in a remarkable improvement of glucose homeostasis and a resolution of diabetes, that typically occurs too fast to be accounted for by weight loss alone. Furthermore, an immediate reduction of blood pressure following laparoscopic gastric bypass has been demonstrated in morbidly obese patients with hypertension as early as one week after the operation. As with the rapid reduction of diabetes, the antihypertensive effect of the procedure might be a consequence of the rearrangement of the gastrointestinal anatomy.

With this study, we want to evaluate the effect of high vs. low sodium intake on blood pressure and system hemodynamics in patients with morbid obesity and to evaluate the impact of laparoscopic gastric bypass on blood pressure, salt sensitivity and body composition in morbidly obese patients. Furthermore, we wants to describe the hemodynamic mechanisms involved in the amelioration of blood pressure during long-term weight loss. Therefore, patients are examined before, 4-6 weeks after and one year after laparoscopic gastric bypass.

Before and one year after the operation, the patients are examined two times; in a five days period of a low dietary sodium consumption and in a five days period of a high sodium consumption respectively. Four-six weeks following the operation, the patients are examined once on their usual diet.

The protocol comprise three sub studies:

1. The effect of high vs low sodium intake on blood pressure and hemodynamics in the morbid obese patient - preoperative study.
2. Effect of gastric bypass surgery on blood pressure, hemodynamics and salt-sensitivity - 1 year follow-up.
3. Effect of gastric bypass surgery on echocardiographic parameters - 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria (cases):

* Caucasians fulfilling the criteria for laparoscopic gastric bypass.
* 12 participants with hypertension, defined as blood pressure > 140/90 and/or use of antihypertensive medication and 12 participants without hypertension.
* Body mass index 40-50 kg/m2

Inclusion Criteria (controls):

* Caucasian.
* No hypertension or use of antihypertensive medication.
* Body mass index < 30 kg/m2

Exclusion Criteria (all):

* Pregnancy
* Chronic obstructive pulmonary disease
* Diabetes mellitus
* Medical treatment with sibutramine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cases are recruited from the Bariatric Clinics at Glostrup Hospital, Koege Hospital and The Private Hospital Hamlet.
  Controls are recruited through public advertisement
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Sodium induced change in 24-hour blood pressure before and one year after laparoscopic gastric bypass. | One year

SECONDARY OUTCOMES:
Echocardiography: Dimensions, systolic and diastolic function before and one year after laparoscopic gastric bypass | One year
Non-invasive hemodynamic measurements (inert gas rebreathing) before and one year after laparoscopic gastric bypass | One year
Body composition: Dexa-scan, plasma volume and extracellular volume before and one year after laparoscopic gastric bypass | One year
Blood samples: MR-proANP, p-glucose, p-insulin | One year

CONTACTS AND LOCATIONS:
Overall Officials: Peter K Bonfils, MD, Principal Investigator — University Hospital Koege; Morten Damgaard, MD, Ph.D., Study Director — Hvidovre Hospital, Copenhagen; Mustafa Taskiran, MD, Ph.D., Study Director — University Hospital Koege; Viggo B Kristiansen, MD, Study Director — Glostrup Hospital, Copenhagen; Knud H Stokholm, MD, Study Director — University Hospital Koege; Niels Gadsboll, MD, DMSc, Study Chair — University Hospital Koege
Locations (1):
- University Hospital Koege, Department of Clinical Physiology and Nuclear Medicine, Koege, Denmark

REFERENCES:
- [Derived] Bonfils PK, Taskiran M, Damgaard M, Goetze JP, Floyd AK, Funch-Jensen P, Kristiansen VB, Stockel M, Bouchelouche PN, Gadsboll N. Roux-en-Y gastric bypass alleviates hypertension and is associated with an increase in mid-regional pro-atrial natriuretic peptide in morbid obese patients. J Hypertens. 2015 Jun;33(6):1215-25. doi: 10.1097/HJH.0000000000000526. PMID 25668345